CLINICAL TRIAL: NCT05348278
Title: Randomized Controlled Trial to Evaluate Efficacy of Urea-based Cream for Prevention of Capecitabine-associated Hand Foot Skin Reactions
Brief Title: Urea Cream Prevention for Capecitabine Associated Hand Foot Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SI790/2021
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Hand-Foot Syndrome
Keywords: hand foot syndrome; capecitabine; urea cream
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention): standard of care including hand and foot care, avoid friction
- urea cream (Experimental): use 10% urea cream apply at both hands and feet twice a day from time of starting capecitabine
  Interventions: Drug: Urea cream

INTERVENTIONS:
Drug: Urea cream — apply 10% urea cream at both hands and feet twice daily
  Other Names: Softcare cream
  Arms: urea cream

SUMMARY:
Hand foot skin reaction (HFS) from capecitabine is one of the most common adverse events from capecitabine. Urea cream has been proved its benefit to prevent HFS from sorafenib. Prior study using urea cream prophylaxis in patients receiving capecitabine was negative. However, result from aformentioned study was reported primarily from result of first cycle capecitabine. Urea cream as a prevention of HFS from capecitabine has been used in clinical practice in Thailand according to expert's opinion. We conducted the study to evaluate wheter the urea cream can prevent HFS or severe HFS.

DETAILED DESCRIPTION:
The patients who is planned to receive capecitabine for at least 3 cycles were enrolled in the study. The patients were randomized to receive 10% urea cream or standard measure. The patients were followed until the end of capecitabine treatment. The patients reported their symptoms of HFS and other adverse events (AE) before starting new cycle of capecitabine. Physician record of HFS and other AE, dose modification of capecitabine and compliance were extracted. We will report incidence of any HFS, > grade 3 HFS, capecitabine interruption or delay or discontinuation and time to develop HFS among both arms. The results of the study will be used for optimal prophylactic measures in patients treated with capecitabine.

ELIGIBILITY:
Inclusion Criteria:

- patients who has plan to receive capecitabine at the dosage of at least 2000 mg/m2 D1-14 every 21 days for at least 3 cycles

Exclusion Criteria:

* preexisting neuropathy which was severe than grade 2
* history of allergy to urea cream
* patients with previous use of capecitabine 2000 mg/m2
* patients who has prior routinely used of urea cream

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
any HFS | from starting capecitabine until 4 week after capecitabine discontinuation
  incidence of any HFS

SECONDARY OUTCOMES:
severe HFS | from starting capecitabine until 4 week after capecitabine discontinuation
  grade 3 or 4 HFS
time to develop severe HFS | from starting capecitabine until 4 week after capecitabine discontinuation
  time for starting capecitabine to time of >grade II HFS reported
capecitabine interruption | from starting capecitabine until 4 week after capecitabine discontinuation
  proportion of patient with capecitabine interruption due to HFS

CONTACTS AND LOCATIONS:
Overall Officials: Suthinee Ithimakin, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of medical oncology, department of medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wongkraisri C, Chusuwanrak K, Laocharoenkeat A, Chularojanamontri L, Nimmannit A, Ithimakin S. Randomized controlled trial on the efficacy of topical urea-based cream in preventing capecitabine-associated hand-foot syndrome. BMC Cancer. 2025 Feb 17;25(1):275. doi: 10.1186/s12885-025-13684-1. PMID 39962445